CLINICAL TRIAL: NCT00148096
Title: Randomised Controlled Trial of Mechanical Heat Recovery Ventilation on Asthma Control of Patients Allergic to the House Dust Mite
Brief Title: Mechanical Heat Recovery Ventilation on House Dust Mite Sensitive Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government); North Lanarkshire Council (Unknown); South Lanarkshire Council (Unknown); North Glasgow Primary Care Trust (Unknown); Vent-axia Ltd (Unknown); Scottish Power (Unknown); Energy Action Scotland (Unknown); Communities Scotland (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CZB/4/47; CSO CZB/4/47 and BO/01/69
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2007-11

CONDITIONS: Asthma
Keywords: asthma; house dust mite; allergy; housing; avoidance; humidity
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Mechanical heat recovery ventilation units installed but not fully functional
  Interventions: Device: Mechanical Heat Recovery Ventilation
- 2 (Active Comparator): Mechanical heat recovery ventilation unit installed and active
  Interventions: Device: Mechanical Heat Recovery Ventilation

INTERVENTIONS:
Device: Mechanical Heat Recovery Ventilation — De-humidification without loss of heat
  Other Names: Ventaxia

SUMMARY:
Asthma has become increasingly common in the UK, demanding our consideration of the cause. Many patients with asthma are allergic to house dust mites, which thrive in modern housing. Improving ventilation in the home has been shown to reduce dust mite levels, by reducing humidity levels. It is hoped that, by removing the dust mites from homes, asthma may improve. In this study, 140 volunteers will have their carpets steam-cleaned and new allergy bedding provided, before a team of architects installs a ventilation system in the loft. Half of the units will be switched on at the beginning of the study. The other half will be switched on in 12 months time, but only the architects know which units are active. The medical team will compare the asthma, and measures of inflammation in the airways, over that year.

It is due for completion in April 2007.

DETAILED DESCRIPTION:
The prevalence of asthma is rising sharply in the UK. The house dust mite is the most common trigger associated with asthma, thriving in the humid microclimate favoured by modern housing. Could this be redressed by investment in improved ventilation in local housing? In a pilot study in North Lanarkshire Council housing stock, we demonstrated that dust mite avoidance, in combination with installation of domestic mechanical heat recovery ventilation (MHRV), could inhibit the re-colonisation of house dust mites by reduction of indoor air humidity. In this second phase, a double blind randomized placebo- controlled trial will test the resultant effect on asthma. It will be complete in November 2006. 140 patients with asthma and house dust mite allergy are being recruited and all will have new bedding, mattress covers and carpets cleaned. All will have MHRV units installed in their home, but only half will be activated, before 12 months of environmental and clinical monitoring. The primary endpoint is morning peak flow rate. Secondary endpoints include symptom scores, spirometry, rates of exacerbations, quality-of-life, and economic evaluations. Demonstration that well ventilated, energy efficient dwellings improve the respiratory health of patients with allergic asthma could be of considerable importance in helping the NHS cope with the commonest chronic disease in Scotland.

ELIGIBILITY:
Inclusion Criteria:

* House dust mite sensitive
* FEV1 greater than 50%
* Symptomatic asthma or 12% reversibility on spirometry or 15%PEFR lability

Exclusion Criteria:

* Multi-storey flat

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 119 (Actual)
Dates: Start 2003-02; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
morning Peak Flow | 1 year

SECONDARY OUTCOMES:
symptom scores | 1 year
exacerbation rates | 1 year
quality of life | 1 year
spirometry | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Prof Neil C Thomson, MD FRCP, Principal Investigator — The University of Glasgow
Locations (1):
- Monklands General Hospital, North Lanarkshire, United Kingdom

REFERENCES:
- See also: Asthma Research Unit website — http://www.gla.ac.uk/departments/immunology/respiratorymedicine/